CLINICAL TRIAL: NCT05031728
Title: Cognitive Processing Therapy for the Treatment of Post-Traumatic Stress Disorder in Syrian Patients
Brief Title: Cognitive Processing Therapy for Syrian Patients With PTSD
Acronym: CPT4Syrians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Amani Safwat Albrazi, Principal Investigator, British University In Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BritishUE20-21
Record Dates: First submitted 2021-08-17; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: Cognitive Processing Therapy (CPT); Posttraumatic stress disorder (PTSD); Syrians
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Patients will be interviewed by a clinician and asked to complete the Clinician-Administered PTSD Scale (CAPS-5), Beck Depression Inventory (BDI-II), Beck Anxiety Inventory (BAI). Assessments will be conducted at baseline, 3-, and 12-months post treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPT Group (Experimental): Cognitive Processing Therapy (CPT) is employed. Each patient will attend 12 individual sessions with the therapist. The sessions will be on the weekly basis. The standard manual of CPT (Resick et al., 2016) is going to be employed.
  Interventions: Behavioral: Cognitive Processing Therapy (CPT)

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy (CPT) — Cognitive processing therapy (CPT) (Resick et al., 2016) which is a specific type of cognitive behavioral therapy that has been effective in reducing symptoms of Post-Traumatic Stress Disorder (PTSD) that may have developed after experiencing a variety of traumatic events including child abuse, emotional abuse, combat, rape war, and natural disasters. CPT helps patients learn how to challenge and modify unhelpful beliefs related to the trauma and emotional pain. In so doing, the client creates a new understanding and conceptualization of the traumatic event so that it reduces its ongoing negative effects on current life.

SUMMARY:
Background: Studies among Syrian refugees showed high prevalence rates of PTSD. The objective of the present study was to investigate the effectiveness of Cognitive Processing Therapy (CPT) in treating patients with posttraumatic stress disorder (PTSD) using a clinical trial. Methods: Data will be obtained through interviewing patients seeking for PTSD treatment. Patients will be interviewed by a clinician and asked to complete the Clinician-Administered PTSD Scale (CAPS-5), Beck Depression Inventory (BDI-II), Beck Anxiety Inventory (BAI). Assessments will be conducted at baseline, 3-, and 12-months posttreatment. The primary outcomes will be the scores of CAPS, BDI-II, and BAI. Results: we predict that CPT will result in greater reductions in CAPS scores.

DETAILED DESCRIPTION:
Although individuals with PTSD experience significant suffering, disability, and a challenging clinical course, there are still significant gaps in the evidence addressing effective treatment options. Therefore, in the current study CPT will determine the effectiveness in treating Syrian patients with PTSD. Current study significantly adds to the existing literature. It is a novel study in Egypt and adds to the literature.

ELIGIBILITY:
Inclusion Criteria Their nationalities are Syrians

* age older than 18 years and younger than 65,
* patients meeting current diagnostic criteria for PTSD as defined in DSM-5
* have a good knowledge of English-language (reading, writing, and comprehension) because all assessments and therapy materials were in English

Exclusion Criteria

* having mental retardation
* having schizophrenia (or any other psychotic disorders).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
assessing change in CAPS-5 scores between three time points | baseline (pre-intervention), posttreatment (immediately after the intervention), 12-months after the intervention
  Clinician-Administered PTSD Scale (CAPS-5; Weathers et al., 2015) is currently the gold- standard assessment for PTSD and is used to assess PTSD's symptoms at pre-intervention, immediately post- intervention, and 12-month after the intervention. This 30-item structured interview was developed by staff at the U.S. Department of Veterans Affairs National Center for PTSD. The interview can generally be administered in 45-60 minutes. Each question in CAPS asks about both the frequency and the severity of each PTSD symptom. These questions are split into categories. Each criterion has several questions, and scores for each criterion are added up at the end. The CAPS-5 has demonstrated strong psychometric properties (Weathers, et al., 2018).

SECONDARY OUTCOMES:
assessing change in Beck Depression Inventory (BDI-II) scores between three time points | baseline (pre-intervention), posttreatment (immediately after the intervention), 12-months after the intervention
  Beck Depression Inventory (BDI-II): was used to evaluate the change in the severity of depressive symptoms between three time points. BDI-II is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression (Beck, et al., 1996). The BDI takes approximately 10 minutes to complete. Depression levels were defined as follows: minimal range = 0- 13, mild depression = 14-19, moderate depression = 20-28, and severe depression = 29- 63.
assessing change in Beck Anxiety Inventory (BAI) scores between three time points | baseline (pre-intervention), posttreatment (immediately after the intervention), 12-months after the intervention
  Beck Anxiety Inventory (BAI): was used to evaluate the change in the severity of anxiety severity between three time points.
  BAI was developed by Dr. Aaron T. Beck and it is a brief measure of anxiety with a focus on somatic symptoms of anxiety such as nervousness, dizziness, inability to relax (Beck et al., 1988). It has a total of 21 items that takes approximately 10-15 minutes to complete. Answers are on a 4-point Likert scale and range from 0 (not at all) to 3 (severely). The values for each item are summed yielding an overall or total score for all 21 symptoms that can range between 0 and 63 points. A total score of 0 - 7 is interpreted as a "Minimal" level of anxiety; 8 - 15 as "Mild"; 16 -25 as "Moderate", and 26 - 63 as "Severe".

CONTACTS AND LOCATIONS:
Overall Officials: Amani S Elbarazi, Ph.D., Principal Investigator — The British University in Egypt
Locations (1):
- The British university in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
individual participant data (IPD) will be available to other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2022
Access Criteria: Direct access to the patients' data will be granted to authorized representatives from the Sponsor and host hospital for monitoring and/or audit of the study to ensure compliance with regulations.